CLINICAL TRIAL: NCT00001714
Title: Magnetization Transfer Quantitation and Characterization for Clinical Scanners
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 980084; 98-CC-0084
Record Dates: First submitted 1999-11-03; First posted 2002-12-10 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-02

CONDITIONS: Healthy
Keywords: MRI; Macromolecules; Magnetization Transfer; Metabolites; Tissue Characterization; Normal Volunteer

SUMMARY:
This project will measure magnetization transfer (MT) parameters on normal subjects using two novel approaches. The first is the investigation of asymmetric MT effects with respect to the zero or on-resonance reference point. The technique measures the difference in MT effect between two symmetrically positioned off-resonance MT pulses in the positive and negative frequency ranges. Prior research with this technique in the kidney show a difference in the macromolecular lineshape that correlates to a specific metabolite. The second approach, utilizing a subset of the acquisitions from the first approach, will test newly developed formulation to calculate the macromolecular fraction, or fraction of proton density that accounts for MT. We foresee these measurements may significantly develop our understanding of MT and introduce diagnostic and quantitative tools to study human tissues.

DETAILED DESCRIPTION:
This project will measure magnetization transfer (MT) parameters on normal subjects using two novel approaches. The first is the investigation of asymmetric MT effects with respect to the zero or on-resonance reference point. The technique measures the difference in MT effect between two symmetrically positioned off-resonance MT pulses in the positive and negative frequency ranges. Prior research with this technique in the kidney show a difference in the macromolecular lineshape that correlates to a specific metabolite. The second approach, utilizing a subset of the acquisitions from the first approach, will test newly developed formulation to calculate the macromolecular fraction, or fraction of proton density that accounts for MT. We foresee these measurements may significantly develop our understanding of MT and introduce diagnostic and quantitative tools to study human tissue.

ELIGIBILITY:
Normal control between the ages of 18 - 70 years of age who are capable of giving informed consent.

Subjects must not have a condition which would preclude their use for technical development (e.g. paralyzed hemidiaphragm, morbid obesity, claustrophobia, etc.).

Subjects must not have a condition which would present unnecessary risks (e.g. pregnancy, surgery of uncertain type, symptoms of pheochromocystoma or insulinoma, etc.).

Lactating women and subjects with hemoglobinopathies, asthma, or renal or hepatic disease will be excluded from studies involving the administration of contrast agents.

Must not have a contraindication to MR scanning such as surgery that involves metal clips or wires which might be expected to concentrate radiofrequency fields or cause tissue damage from twisting in a magnetic field. Examples include: aneurysm clip; implanted neural stimulator; implanted cardiac pacemaker or autodefibrillator; cochlear implant; ocular foreign body (e.g. metal shavings); insulin pump.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1998-03; Study Completion 2001-07

CONTACTS AND LOCATIONS:
Locations (1):
- Warren G. Magnuson Clinical Center (CC), Bethesda, Maryland, United States

REFERENCES:
- [Background] Bottomley PA, Foster TH, Argersinger RE, Pfeifer LM. A review of normal tissue hydrogen NMR relaxation times and relaxation mechanisms from 1-100 MHz: dependence on tissue type, NMR frequency, temperature, species, excision, and age. Med Phys. 1984 Jul-Aug;11(4):425-48. doi: 10.1118/1.595535. PMID 6482839
- [Background] Wolff SD, Balaban RS. Magnetization transfer contrast (MTC) and tissue water proton relaxation in vivo. Magn Reson Med. 1989 Apr;10(1):135-44. doi: 10.1002/mrm.1910100113. PMID 2547135
- [Background] Wolff SD, Balaban RS. Magnetization transfer imaging: practical aspects and clinical applications. Radiology. 1994 Sep;192(3):593-9. doi: 10.1148/radiology.192.3.8058919. No abstract available.